CLINICAL TRIAL: NCT05435677
Title: A Study Investigating the Pharmacokinetic Properties of a Single Dose of IcoSema Compared With Insulin Icodec and Semaglutide Given Separately in Chinese Participants With Type 2 Diabetes
Brief Title: A Research Study to Look at How Insulin Icodec and Semaglutide Work in the Body of People From China With Type 2 Diabetes When Given Alone or Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1535-4710; U1111-1262-1959 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): All participants will get each of the 3 medicines at 3 different timepoints IcoSema - insulin icodec - semaglutide, separated by a 1-4-week wash-out period. The study will last for about 19 to 26 weeks.
  Interventions: Drug: IcoSema; Drug: insulin icodec; Drug: semaglutide
- Sequence 2 (Experimental): All participants will get each of the 3 medicines at 3 different timepoints IcoSema- semaglutide . insulin icodec, separated by a 1-4-week wash-out period. The study will last for about 19 to 26 weeks.
  Interventions: Drug: IcoSema; Drug: insulin icodec; Drug: semaglutide
- Sequence 3 (Experimental): All participants will get each of the 3 medicines at 3 different timepoints insulin icodec- IcoSema- semaglutide, separated by a 1-4-week wash-out period. The study will last for about 19 to 26 weeks.
  Interventions: Drug: IcoSema; Drug: insulin icodec; Drug: semaglutide
- Sequence 4 (Experimental): All participants will get each of the 3 medicines at 3 different timepoints insulin icodec- semaglutide - IcoSema separated by a 1-4-week wash-out period. The study will last for about 19 to 26 weeks.
  Interventions: Drug: IcoSema; Drug: insulin icodec; Drug: semaglutide
- Sequence 5 (Experimental): All participants will get each of the 3 medicines at 3 different timepoints semaglutide - IcoSema - insulin icodec, separated by a 1-4-week wash-out period. The study will last for about 19 to 26 weeks.
  Interventions: Drug: IcoSema; Drug: insulin icodec; Drug: semaglutide
- Sequence 6 (Experimental): All participants will get each of the 3 medicines at 3 different timepoints semaglutide - insulin icodec - IcoSema, separated by a 1-4-week wash-out period. The study will last for about 19 to 26 weeks.
  Interventions: Drug: IcoSema; Drug: insulin icodec; Drug: semaglutide

INTERVENTIONS:
Drug: IcoSema — One single dose of IcoSema administered subcutaneously, S.c. into the left thigh
Drug: insulin icodec — One single dose of insulin icodec administered subcutaneously, S.c. into the left thigh
Drug: semaglutide — One single dose of semaglutide administered subcutaneously, S.c. into the left thigh

SUMMARY:
This study will look at a new medicine, called IcoSema, for treatment of type 2 diabetes.

IcoSema is a combination of a new insulin, called insulin icodec, and a GLP-1 receptor analogue, called semaglutide.

Insulin icodec is a possible new medicine. That means that the medicine has not yet been approved by the authorities. Semaglutide is a medicine already approved by the authorities in the EU, USA, China and Japan.

The study will look at the way insulin icodec and semaglutide reach and stay in participants blood after injection when given together as IcoSema or alone as insulin icodec and semaglutide.

Participants will get each of the 3 medicines (IcoSema, insulin icodec and semaglutide) at 3 different timepoints:

The order in which participants get them is decided by chance. Participants will get the 3 medicines as an injection under the skin in the thigh. The injections will be done by study staff. The time between injections is 6 to 9 weeks.

The study will last for about 19 to 26 weeks. Participants will have 31 or 32 visits to the clinic. 3 of the visits will be in-house visits, meaning that participants will stay at the clinic for 5 or 6 days (4 or 5 nights).

Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female
* Aged 18-64 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of screening
* Body mass index between 18.5 and 34.9 kg/m^2 (both inclusive)
* Body weight greater than or equal to 50 kg
* HbA1c (glycated haemoglobin) below or equal to 9.0% (75 mmol/mol)
* Insulin naïve. However, short-term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes
* Stable daily dose(s) including any of the following anti-diabetic drug(s)/regimen within 45 days prior to the day of screening:

  * Any metformin formulation
  * DPP-4 (dipeptidyl peptidase-4) inhibitors (participants are not allowed to participate in the study if they are treated with DPP-4 inhibitors as monotherapy)
  * SGLT2 (sodium-glucose linked transporter 2) inhibitors
  * Alpha-glucosidase inhibitors
  * Oral combination products (for the allowed individual oral antidiabetic drugs)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive method
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event within the past 180 days) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis within the past 180 days prior to the day of screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
AUCIco,0-tz:Area under the serum insulin icodec concentration-time curve after a single dose | From 0 hours to tz hours after IMP administration (day 1) where tz is the time of the last quantifiable concentration
  Measured in hours*pmol/L
Dose-normalised AUCSema,0-tz: Area under the plasma semaglutide concentration-time curve after a single dose divided by dose | From 0 hours to tz hours after IMP administration (day 1) where tz is the time of the last quantifiable concentration
  Measured in (hours*nmol/L)/mg

SECONDARY OUTCOMES:
AUCIco,0-inf: Area under the serum insulin icodec concentration-time curve after a single dose | From 0 hours to infinity after IMP administration (day 1)
  Measured in hours*pmol/L
Cmax,Ico: Maximum observed serum insulin icodec concentration after a single dose | From 0 hours until last measurement time after IMP administration (day 1)
  Measured in pmol/L
tmax,Ico: Time to maximum observed serum insulin icodec concentration after a single dose | From 0 hours until last measurement time after IMP administration (day 1)
  Measured in hours
t1/2,Ico: Terminal half-life for insulin icodec after a single dose | Terminal part of the serum insulin icodec concentration-time curve where the curve is well approximated by a straight line on logarithmic scale after IMP administration (day 1)
  Measured in hours
Dose-normalised AUCSema,0-inf: Area under the plasma semaglutide concentration-time curve after a single dose divided by dose | From 0 hours to infinity after IMP administration (day 1)
  Measured in (hours*nmol/L)/mg
Dose-normalised Cmax,Sema: Maximum observed plasma semaglutide concentration after a single dose divided by dose | From 0 hours until last measurement time after IMP administration (day 1)
  Measured in (nmol/L)/mg
tmax,Sema: Time to maximum observed plasma semaglutide concentration after a single dose | From 0 hours until last measurement time after IMP administration (day 1)
  Measured in hours
t1/2,Sema: Terminal half-life for semaglutide after a single dose | Terminal part of the plasma semaglutide concentration-time curve where the curve is well approximated by a straight line on logarithmic scale after IMP administration (day 1)
  Measured in hours
Adverse events | From IMP administration (day 1) to end of follow-up for each treatment period (day 36)
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Peking University Third Hospital, Northern branch-Phase I, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Wang F, Luan Z, Maltesen R, Reenberg AT, Westergaard L, Liu D. Pharmacokinetic Characteristics of a Once-Weekly Combination Therapy of Insulin Icodec and Semaglutide Versus Its Separate Components in Chinese Individuals with Type 2 Diabetes. Diabetes Ther. 2025 Nov;16(11):2213-2225. doi: 10.1007/s13300-025-01803-x. Epub 2025 Oct 6. PMID 41051695